CLINICAL TRIAL: NCT04125121
Title: Neuroplasticity Induced by General Anaesthesia
Acronym: DANA1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Signe Sloth Madsen (Other)
Responsible Party: Sponsor-Investigator, Signe Sloth Madsen, Principal Investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-18028925
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Healthy Volunteers; General Anaesthesia; Neuroplasticity
Keywords: Neuroplasticity; Neuroplastic changes; General anaesthesia; Magnetic resonance imaging; Sevoflurane; Propofol; Healthy volunteers; Consciousness; Cognitive; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Randomisation to one of two options in session 1: sevoflurane or propofol. In session 2, the remaining option is administered.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants will not be present during randomisation. The participants will be anaesthetised when the investigational drug (maintenance anaesthetic) is administered, and will thus not be aware what type of anaesthesia is administered in which (otherwise identical) session.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane-Propofol (Active Comparator): Session one: Sevoflurane as maintenance anaesthetic during general anaesthesia.
  Session two: Propofol as maintenance anaesthetic during general anaesthesia.
  Interventions: Drug: Sevoflurane-propofol
- Propofol-Sevoflurane (Active Comparator): Session one: Propofol as maintenance anaesthetic during general anaesthesia.
  Session two: Sevoflurane as maintenance anaesthetic during general anaesthesia.
  Interventions: Drug: Sevoflurane-propofol

INTERVENTIONS:
Drug: Sevoflurane-propofol — General anaesthesia with a maintenance phase of two hours duration with either sevoflurane or propofol.
  Other Names: Propofol-sevoflurane

SUMMARY:
The aim of this study is to use magnetic resonance imaging to explore and compare possible de novo neuroplastic changes induced by the isolated effects of the hypnotic agents sevoflurane and propofol, respectively. In addition, to explore possible associations between neuroplastic changes and clinical and/or biochemical outcomes. It is a randomised, cross-over, single blinded clinical study. N = 30. Female:male ratio 1:1.

DETAILED DESCRIPTION:
Background

In the perioperative period, severe changes can be observed in the endocrine, immune, and nervous system. These changes are called the surgical stress response. Clinically, this can be observed as increased pain response and disturbances in the circadian rhythm, memory, cognitive and executive functions, and may lead to post-operative delirium. The post-operative cognitive dysfunction is associated with increased mortality and risk of prematurely leaving occupation. Post-operative delirium with fluctuating levels of attention and consciousness is a serious condition associated with poor outcome, including longer hospitalisation and increased early mortality.

General anaesthesia may contribute to the surgical stress response. Some data indicate that general anaesthesia per se can cause alterations and disturbances in the brain such as sleep and circadian disturbances. Recent evidence suggests that anaesthetic agents may impair neurogenesis and cause memory impairment. In addition, inhalation anaesthesia may result in more cerebral disturbances compared to total intravenous anaesthesia (TIVA). In this study, we will isolate the effects of the two primary hypnotic agents used in general anaesthesia, sevoflurane and propofol, without the interactions and confounders of polypharmacy and varying levels of disease among a surgical population.

Materials

The study consists of two study sessions. In each study session magnetic resonance imaging (MRI) scans will be obtained before and after general anaesthesia, and in addition after one and eight days.

The following imaging modalities will be employed: (i) T1-weighted 3D anatomy (T1w3D), (ii) Diffusion Tensor Imaging (DTI), (iii) resting state functional MRI (rsfMRI). The MRI scans will be supplemented with cognitive testing, sleep evaluation and blood sampling. Thus, the set-up for each volunteer will be:

Session one:

Day 0: MRI 1, cognitive testing, questionnaires, and blood sampling. General anaesthesia (maintenance phase with sevoflurane OR propofol according to randomisation), and post-anaesthesia care. MRI 2 and repeated cognitive testing, questionnaires, and blood sampling.

Day +1: MRI 3, cognitive testing, questionnaires, and blood sampling.

Day +8: MRI 4, cognitive testing, and questionnaires.

Session two: Identical to session one, except the volunteer will receive the remaining type of general anaesthesia (sevoflurane or propofol, opposite to session one).

Data evaluation will be conducted with assessor blinded to anaesthesia type.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤35.
* Healthy individual.
* BMI ≥18 kg/m2 and ≤30kg/m2.
* Normal electrocardiogram (ECG).
* Normal physical examination, including neurological examination, auscultation of the heart and lungs, and measurement of blood pressure and pulse.
* American Society of Anaesthesiologists (ASA) class 1.
* Mallampati I-II and simplified airway risk index (SARI) 0-2 (i.e. no indication of difficult intubation). See appendix for details.
* Right-handed.
* Female participants must use safe contraceptives (hormonal or mechanical, including intrauterine devices).
* Speaks and understand Danish.
* Provides oral and written informed consent.

Exclusion Criteria:

* Contraindications to MRI.
* Left-handedness or ambidexterity.
* History of complications to general anaesthesia, including malignant hyperthermia.
* Family history of malignant hyperthermia.
* Known incident of malignant hyperthermia or any unexplained complication to general anaesthesia among close relatives.
* Allergy to any kind of medication or material to which the volunteer could be exposed during this study.
* History of serious illness.
* History of cancer, immune disease, autoimmune disease, chronic pain or neurological / psychiatric illness.
* Major trauma or head trauma with any symptoms present at the time of inclusion.
* Surgery less than six weeks prior to the study period.
* Infection (with fever) less than two weeks prior to or during the study sessions.
* Daily use of any medication (not counting contraceptives).
* Consumed anti-depressants during the last 30 days before study days.
* Weakly intake of >21 (for females >14) units of alcohol.
* Heavy intake of caffeine (> 5 cups/day).
* Smoking during the last 30 days before study days.
* Substance abuse (assessed by the investigator).
* Pregnancy
* Reflux or dyspepsia.
* Poor dental status or oral health.
* Expected or suspected difficult airway.
* Declines receiving information regarding accidental pathological findings during MRI scans of the brain.
* Cannot cooperate to tests.
* Otherwise judged unfit for participation by the investigator.

Exclusion Criteria during the study:

* Any of the above-mentioned exclusion criteria.
* Major trauma or head trauma during the study period.
* Surgery during the study period.
* Infection (with fever) during the study period.
* Consumption of more than 3 units of alcohol within 24 hours before each study day (intervention day or MRI scan day)
* Consumed analgesics within 3 days before each study day
* Consumed anti-histamines less than 48 hours before each study day
* Intake of caffeine 12 h prior to each study day
* Smoking

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
Changes in T1w3D | 8 days
  Volume and morphology of selected brain regions and anatomical structures as recorded by T1w3D anatomy MRI.
Changes in DTI | 8 days
  White matter microstructure as measured using Diffusion Tensor Imaging (DTI)

SECONDARY OUTCOMES:
Changes in rsfMRI | 8 days
  Differences in resting state functional MRI induced by general anaesthesia
Changes in fatigue | 8 days
  Differences in severity and characteristics of fatigue related to general anaesthesia, as measured by Multidimensional Fatigue Inventory (MFI-20, a scale of 0-5 in each of 20 questions, with higher scores indicating more fatigue).
Cognitive performance | 8 days
  Changes in cognitive function related to general anaesthesia, measured with a combination of Test of Attentional Performance, Paced Auditory Serial Addition Test and Conners Continuous Performance Test.

CONTACTS AND LOCATIONS:
Overall Officials: Signe Madsen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Department of Neuroanaesthesiology, Glostrup Municipality, Capital Region
  - Functional Imaging Unit, Department for Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet Glostrup, Glostrup Municipality, Capital Region

IPD SHARING:
Plan to Share IPD: No
The responsible investigators will consider data sharing, considered compliance with General Data Protection Regulation (GDPR) regulations and data sharing agreement.

REFERENCES:
- [Background] Miller G. Miller's Anesthesia. 2015 ed. Philadelphia: Elsevier Saunders; 2015.
- [Background] Campagna JA, Miller KW, Forman SA. Mechanisms of actions of inhaled anesthetics. N Engl J Med. 2003 May 22;348(21):2110-24. doi: 10.1056/NEJMra021261. No abstract available. PMID 12761368
- [Background] Ishizawa Y. Mechanisms of anesthetic actions and the brain. J Anesth. 2007;21(2):187-99. doi: 10.1007/s00540-006-0482-x. Epub 2007 May 30. PMID 17458649
- [Background] Vanlersberghe C, Camu F. Propofol. Handb Exp Pharmacol. 2008;(182):227-52. doi: 10.1007/978-3-540-74806-9_11. PMID 18175094
- [Background] Dunnet JM, Prys-Roberts C, Holland DE, Browne BL. Propofol infusion and the suppression of consciousness: dose requirements to induce loss of consciousness and to suppress response to noxious and non-noxious stimuli. Br J Anaesth. 1994 Jan;72(1):29-34. doi: 10.1093/bja/72.1.29. PMID 8110545
- [Background] Forrest FC, Tooley MA, Saunders PR, Prys-Roberts C. Propofol infusion and the suppression of consciousness: the EEG and dose requirements. Br J Anaesth. 1994 Jan;72(1):35-41. doi: 10.1093/bja/72.1.35. PMID 8110547
- [Background] Casati A, Fanelli G, Casaletti E, Colnaghi E, Cedrati V, Torri G. Clinical assessment of target-controlled infusion of propofol during monitored anesthesia care. Can J Anaesth. 1999 Mar;46(3):235-9. doi: 10.1007/BF03012602. PMID 10210047
- [Background] Sukhotinsky I, Zalkind V, Lu J, Hopkins DA, Saper CB, Devor M. Neural pathways associated with loss of consciousness caused by intracerebral microinjection of GABA A-active anesthetics. Eur J Neurosci. 2007 Mar;25(5):1417-36. doi: 10.1111/j.1460-9568.2007.05399.x. PMID 17425568
- [Background] Miller G. What is the biological basis of consciousness? Science. 2005 Jul 1;309(5731):79. doi: 10.1126/science.309.5731.79. No abstract available. PMID 15994525
- [Background] Schneider G, Kochs EF. The search for structures and mechanisms controlling anesthesia-induced unconsciousness. Anesthesiology. 2007 Aug;107(2):195-8. doi: 10.1097/01.anes.0000271869.27956.d1. No abstract available. PMID 17667560
- [Background] Brown EN, Lydic R, Schiff ND. General anesthesia, sleep, and coma. N Engl J Med. 2010 Dec 30;363(27):2638-50. doi: 10.1056/NEJMra0808281. No abstract available. PMID 21190458
- [Background] Herling SF, Dreijer B, Wrist Lam G, Thomsen T, Moller AM. Total intravenous anaesthesia versus inhalational anaesthesia for adults undergoing transabdominal robotic assisted laparoscopic surgery. Cochrane Database Syst Rev. 2017 Apr 4;4(4):CD011387. doi: 10.1002/14651858.CD011387.pub2. PMID 28374886
- [Background] Steinmetz J, Christensen KB, Lund T, Lohse N, Rasmussen LS; ISPOCD Group. Long-term consequences of postoperative cognitive dysfunction. Anesthesiology. 2009 Mar;110(3):548-55. doi: 10.1097/ALN.0b013e318195b569. PMID 19225398
- [Background] Witlox J, Eurelings LS, de Jonghe JF, Kalisvaart KJ, Eikelenboom P, van Gool WA. Delirium in elderly patients and the risk of postdischarge mortality, institutionalization, and dementia: a meta-analysis. JAMA. 2010 Jul 28;304(4):443-51. doi: 10.1001/jama.2010.1013. PMID 20664045
- [Background] Inouye SK, Marcantonio ER, Kosar CM, Tommet D, Schmitt EM, Travison TG, Saczynski JS, Ngo LH, Alsop DC, Jones RN. The short-term and long-term relationship between delirium and cognitive trajectory in older surgical patients. Alzheimers Dement. 2016 Jul;12(7):766-75. doi: 10.1016/j.jalz.2016.03.005. Epub 2016 Apr 18. PMID 27103261
- [Background] Newman MF, Grocott HP, Mathew JP, White WD, Landolfo K, Reves JG, Laskowitz DT, Mark DB, Blumenthal JA; Neurologic Outcome Research Group and the Cardiothoracic Anesthesia Research Endeavors (CARE) Investigators of the Duke Heart Center. Report of the substudy assessing the impact of neurocognitive function on quality of life 5 years after cardiac surgery. Stroke. 2001 Dec 1;32(12):2874-81. doi: 10.1161/hs1201.099803. PMID 11739990
- [Background] Strom C, Rasmussen LS, Sieber FE. Should general anaesthesia be avoided in the elderly? Anaesthesia. 2014 Jan;69 Suppl 1(Suppl 1):35-44. doi: 10.1111/anae.12493. PMID 24303859
- [Background] Davis N, Lee M, Lin AY, Lynch L, Monteleone M, Falzon L, Ispahany N, Lei S. Postoperative cognitive function following general versus regional anesthesia: a systematic review. J Neurosurg Anesthesiol. 2014 Oct;26(4):369-76. doi: 10.1097/ANA.0000000000000120. PMID 25144505
- [Background] Lindqvist M, Schening A, Granstrom A, Bjorne H, Jakobsson JG. Cognitive recovery after ambulatory anaesthesia based on desflurane or propofol: a prospective randomised study. Acta Anaesthesiol Scand. 2014 Oct;58(9):1111-20. doi: 10.1111/aas.12381. Epub 2014 Aug 6. PMID 25100438
- [Background] Larsen B, Seitz A, Larsen R. Recovery of cognitive function after remifentanil-propofol anesthesia: a comparison with desflurane and sevoflurane anesthesia. Anesth Analg. 2000 Jan;90(1):168-74. doi: 10.1097/00000539-200001000-00035. PMID 10624999
- [Background] Jevtovic-Todorovic V, Absalom AR, Blomgren K, Brambrink A, Crosby G, Culley DJ, Fiskum G, Giffard RG, Herold KF, Loepke AW, Ma D, Orser BA, Planel E, Slikker W Jr, Soriano SG, Stratmann G, Vutskits L, Xie Z, Hemmings HC Jr. Anaesthetic neurotoxicity and neuroplasticity: an expert group report and statement based on the BJA Salzburg Seminar. Br J Anaesth. 2013 Aug;111(2):143-51. doi: 10.1093/bja/aet177. Epub 2013 May 30. PMID 23722106
- [Background] Schilling T, Kozian A, Senturk M, Huth C, Reinhold A, Hedenstierna G, Hachenberg T. Effects of volatile and intravenous anesthesia on the alveolar and systemic inflammatory response in thoracic surgical patients. Anesthesiology. 2011 Jul;115(1):65-74. doi: 10.1097/ALN.0b013e318214b9de. PMID 21399490
- [Background] Braz MG, Braz LG, Braz JR, Pierine DT, Correa CR, Ferreira AL, Carvalho LR, Yeum KJ, Salvadori DM. Comparison of oxidative stress in ASA physical status I patients scheduled for minimally invasive surgery under balanced or intravenous anesthesia. Minerva Anestesiol. 2013 Sep;79(9):1030-8. Epub 2013 Apr 18. PMID 23598734
- [Background] Crozier TA, Muller JE, Quittkat D, Sydow M, Wuttke W, Kettler D. Effect of anaesthesia on the cytokine responses to abdominal surgery. Br J Anaesth. 1994 Mar;72(3):280-5. doi: 10.1093/bja/72.3.280. PMID 8130044
- [Background] Bartal I, Melamed R, Greenfeld K, Atzil S, Glasner A, Domankevich V, Naor R, Beilin B, Yardeni IZ, Ben-Eliyahu S. Immune perturbations in patients along the perioperative period: alterations in cell surface markers and leukocyte subtypes before and after surgery. Brain Behav Immun. 2010 Mar;24(3):376-86. doi: 10.1016/j.bbi.2009.02.010. Epub 2009 Feb 28. PMID 19254757
- [Background] Ashburner J, Friston KJ. Voxel-based morphometry--the methods. Neuroimage. 2000 Jun;11(6 Pt 1):805-21. doi: 10.1006/nimg.2000.0582. PMID 10860804
- [Background] Ogawa S, Lee TM, Nayak AS, Glynn P. Oxygenation-sensitive contrast in magnetic resonance image of rodent brain at high magnetic fields. Magn Reson Med. 1990 Apr;14(1):68-78. doi: 10.1002/mrm.1910140108. PMID 2161986
- [Background] Brooks J, Tracey I. From nociception to pain perception: imaging the spinal and supraspinal pathways. J Anat. 2005 Jul;207(1):19-33. doi: 10.1111/j.1469-7580.2005.00428.x. PMID 16011543
- [Background] van den Heuvel MP, Hulshoff Pol HE. Exploring the brain network: a review on resting-state fMRI functional connectivity. Eur Neuropsychopharmacol. 2010 Aug;20(8):519-34. doi: 10.1016/j.euroneuro.2010.03.008. Epub 2010 May 14. PMID 20471808
- [Background] Pryor KO, Root JC, Mehta M, Stern E, Pan H, Veselis RA, Silbersweig DA. Effect of propofol on the medial temporal lobe emotional memory system: a functional magnetic resonance imaging study in human subjects. Br J Anaesth. 2015 Jul;115 Suppl 1(Suppl 1):i104-i113. doi: 10.1093/bja/aev038. PMID 26174294
- [Background] Quan X, Yi J, Ye TH, Tian SY, Zou L, Yu XR, Huang YG. Propofol and memory: a study using a process dissociation procedure and functional magnetic resonance imaging. Anaesthesia. 2013 Apr;68(4):391-9. doi: 10.1111/anae.12147. PMID 23488834
- [Background] Mhuircheartaigh RN, Rosenorn-Lanng D, Wise R, Jbabdi S, Rogers R, Tracey I. Cortical and subcortical connectivity changes during decreasing levels of consciousness in humans: a functional magnetic resonance imaging study using propofol. J Neurosci. 2010 Jul 7;30(27):9095-102. doi: 10.1523/JNEUROSCI.5516-09.2010. PMID 20610743
- [Background] Ni Mhuircheartaigh R, Warnaby C, Rogers R, Jbabdi S, Tracey I. Slow-wave activity saturation and thalamocortical isolation during propofol anesthesia in humans. Sci Transl Med. 2013 Oct 23;5(208):208ra148. doi: 10.1126/scitranslmed.3006007. PMID 24154602
- [Background] Bonhomme V, Fiset P, Meuret P, Backman S, Plourde G, Paus T, Bushnell MC, Evans AC. Propofol anesthesia and cerebral blood flow changes elicited by vibrotactile stimulation: a positron emission tomography study. J Neurophysiol. 2001 Mar;85(3):1299-308. doi: 10.1152/jn.2001.85.3.1299. PMID 11247998
- [Background] Pedersen JL, Lilleso J, Hammer NA, Werner MU, Holte K, Lacouture PG, Kehlet H. Thiopental and propofol affect different regions of the brain at similar pharmacologic effects. Anesth Analg. 2004 Aug;99(2):912-918. doi: 10.1213/01.ANE.0000131971.92180.DF. PMID 15271714
- [Background] Hofbauer RK, Fiset P, Plourde G, Backman SB, Bushnell MC. Dose-dependent effects of propofol on the central processing of thermal pain. Anesthesiology. 2004 Feb;100(2):386-94. doi: 10.1097/00000542-200402000-00031. PMID 14739816
- [Background] Sun X, Zhang H, Gao C, Zhang G, Xu L, Lv M, Chai W. Imaging the effects of propofol on human cerebral glucose metabolism using positron emission tomography. J Int Med Res. 2008 Nov-Dec;36(6):1305-10. doi: 10.1177/147323000803600618. PMID 19094440
- [Background] Schlunzen L, Juul N, Hansen KV, Cold GE. Regional cerebral blood flow and glucose metabolism during propofol anaesthesia in healthy subjects studied with positron emission tomography. Acta Anaesthesiol Scand. 2012 Feb;56(2):248-55. doi: 10.1111/j.1399-6576.2011.02561.x. Epub 2011 Oct 19. PMID 22091956
- [Background] Ramani R, Qiu M, Constable RT. Sevoflurane 0.25 MAC preferentially affects higher order association areas: a functional magnetic resonance imaging study in volunteers. Anesth Analg. 2007 Sep;105(3):648-55. doi: 10.1213/01.ane.0000277496.12747.29. PMID 17717218
- [Background] Qiu M, Ramani R, Swetye M, Rajeevan N, Constable RT. Anesthetic effects on regional CBF, BOLD, and the coupling between task-induced changes in CBF and BOLD: an fMRI study in normal human subjects. Magn Reson Med. 2008 Oct;60(4):987-96. doi: 10.1002/mrm.21759. PMID 18816821
- [Background] Lorenz IH, Kolbitsch C, Hormann C, Schocke M, Felber S, Zschiegner F, Hinteregger M, Kremser C, Pfeiffer KP, Benzer A. Subanesthetic concentration of sevoflurane increases regional cerebral blood flow more, but regional cerebral blood volume less, than subanesthetic concentration of isoflurane in human volunteers. J Neurosurg Anesthesiol. 2001 Oct;13(4):288-95. doi: 10.1097/00008506-200110000-00002. PMID 11733659
- [Background] Peltier SJ, Kerssens C, Hamann SB, Sebel PS, Byas-Smith M, Hu X. Functional connectivity changes with concentration of sevoflurane anesthesia. Neuroreport. 2005 Feb 28;16(3):285-8. doi: 10.1097/00001756-200502280-00017. PMID 15706237
- [Background] Kaisti KK, Langsjo JW, Aalto S, Oikonen V, Sipila H, Teras M, Hinkka S, Metsahonkala L, Scheinin H. Effects of sevoflurane, propofol, and adjunct nitrous oxide on regional cerebral blood flow, oxygen consumption, and blood volume in humans. Anesthesiology. 2003 Sep;99(3):603-13. doi: 10.1097/00000542-200309000-00015. PMID 12960544
- [Background] Smith I, Kranke P, Murat I, Smith A, O'Sullivan G, Soreide E, Spies C, in't Veld B; European Society of Anaesthesiology. Perioperative fasting in adults and children: guidelines from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2011 Aug;28(8):556-69. doi: 10.1097/EJA.0b013e3283495ba1. PMID 21712716
- [Background] Struys MM, Sahinovic M, Lichtenbelt BJ, Vereecke HE, Absalom AR. Optimizing intravenous drug administration by applying pharmacokinetic/pharmacodynamic concepts. Br J Anaesth. 2011 Jul;107(1):38-47. doi: 10.1093/bja/aer108. Epub 2011 May 30. PMID 21624964
- [Background] Sahinovic MM, Absalom AR, Struys MM. Administration and monitoring of intravenous anesthetics. Curr Opin Anaesthesiol. 2010 Dec;23(6):734-40. doi: 10.1097/ACO.0b013e3283404579. PMID 21037476
- [Background] Masui K, Upton RN, Doufas AG, Coetzee JF, Kazama T, Mortier EP, Struys MM. The performance of compartmental and physiologically based recirculatory pharmacokinetic models for propofol: a comparison using bolus, continuous, and target-controlled infusion data. Anesth Analg. 2010 Aug;111(2):368-79. doi: 10.1213/ANE.0b013e3181bdcf5b. Epub 2009 Oct 27. PMID 19861357
- [Background] Vestergaard MB, Lindberg U, Aachmann-Andersen NJ, Lisbjerg K, Christensen SJ, Rasmussen P, Olsen NV, Law I, Larsson HB, Henriksen OM. Comparison of global cerebral blood flow measured by phase-contrast mapping MRI with 15 O-H2 O positron emission tomography. J Magn Reson Imaging. 2017 Mar;45(3):692-699. doi: 10.1002/jmri.25442. Epub 2016 Sep 13. PMID 27619317
- [Background] American Society of Anesthesiologists Task Force on Postanesthetic Care. Practice guidelines for postanesthetic care: a report by the American Society of Anesthesiologists Task Force on Postanesthetic Care. Anesthesiology. 2002 Mar;96(3):742-52. doi: 10.1097/00000542-200203000-00033. No abstract available. PMID 11873052
- [Background] Jain V, Langham MC, Wehrli FW. MRI estimation of global brain oxygen consumption rate. J Cereb Blood Flow Metab. 2010 Sep;30(9):1598-607. doi: 10.1038/jcbfm.2010.49. Epub 2010 Apr 21. PMID 20407465
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775
- [Background] Granert O, Peller M, Gaser C, Groppa S, Hallett M, Knutzen A, Deuschl G, Zeuner KE, Siebner HR. Manual activity shapes structure and function in contralateral human motor hand area. Neuroimage. 2011 Jan 1;54(1):32-41. doi: 10.1016/j.neuroimage.2010.08.013. Epub 2010 Aug 12. PMID 20708692
- [Background] Martensson J, Eriksson J, Bodammer NC, Lindgren M, Johansson M, Nyberg L, Lovden M. Growth of language-related brain areas after foreign language learning. Neuroimage. 2012 Oct 15;63(1):240-4. doi: 10.1016/j.neuroimage.2012.06.043. Epub 2012 Jun 29. PMID 22750568
- [Background] Kuhn S, Gleich T, Lorenz RC, Lindenberger U, Gallinat J. Playing Super Mario induces structural brain plasticity: gray matter changes resulting from training with a commercial video game. Mol Psychiatry. 2014 Feb;19(2):265-71. doi: 10.1038/mp.2013.120. Epub 2013 Oct 29. PMID 24166407
- [Background] Chen MH, Liao Y, Rong PF, Hu R, Lin GX, Ouyang W. Hippocampal volume reduction in elderly patients at risk for postoperative cognitive dysfunction. J Anesth. 2013 Aug;27(4):487-92. doi: 10.1007/s00540-012-1548-6. Epub 2013 Jan 31. PMID 23371369
- [Background] Bigler ED, Blatter DD, Anderson CV, Johnson SC, Gale SD, Hopkins RO, Burnett B. Hippocampal volume in normal aging and traumatic brain injury. AJNR Am J Neuroradiol. 1997 Jan;18(1):11-23. PMID 9010515
- [Background] Sagi Y, Tavor I, Hofstetter S, Tzur-Moryosef S, Blumenfeld-Katzir T, Assaf Y. Learning in the fast lane: new insights into neuroplasticity. Neuron. 2012 Mar 22;73(6):1195-203. doi: 10.1016/j.neuron.2012.01.025. Epub 2012 Mar 21. PMID 22445346
- [Background] Boveroux P, Vanhaudenhuyse A, Bruno MA, Noirhomme Q, Lauwick S, Luxen A, Degueldre C, Plenevaux A, Schnakers C, Phillips C, Brichant JF, Bonhomme V, Maquet P, Greicius MD, Laureys S, Boly M. Breakdown of within- and between-network resting state functional magnetic resonance imaging connectivity during propofol-induced loss of consciousness. Anesthesiology. 2010 Nov;113(5):1038-53. doi: 10.1097/ALN.0b013e3181f697f5. PMID 20885292
- [Background] Thirion B, Dodel S, Poline JB. Detection of signal synchronizations in resting-state fMRI datasets. Neuroimage. 2006 Jan 1;29(1):321-7. doi: 10.1016/j.neuroimage.2005.06.054. Epub 2005 Aug 29. PMID 16129624
- [Background] Desmond JE, Glover GH. Estimating sample size in functional MRI (fMRI) neuroimaging studies: statistical power analyses. J Neurosci Methods. 2002 Aug 30;118(2):115-28. doi: 10.1016/s0165-0270(02)00121-8. PMID 12204303
- [Background] Steinmetz LRaJ. Anæstesi. 4 ed. Denmark: FADL's Forlag; 2014 24. marts 2014.
- [Background] Warner ME, Benenfeld SM, Warner MA, Schroeder DR, Maxson PM. Perianesthetic dental injuries: frequency, outcomes, and risk factors. Anesthesiology. 1999 May;90(5):1302-5. doi: 10.1097/00000542-199905000-00013. PMID 10319777
- [Background] Editors ICoMJ. Recommendations for the Conduct, Reporting, Editing, and Publication of Scholarly Work in Medical Journals [Web page, recommandation]. Online: Annals of Internal Medicine / American College of Physicians.; 1978 (updated 2017) [cited 2018 20.03.2018]. Available from: http://www.icmje.org/recommendations/.
- [Background] Universities WgsubtMoHEaSatoD. The Danish Code of Conduct for Research Integrity [Code of conduct]. Online (www.ufm.dk): Danish Ministry of Higher Education and Science; 2014 [updated June 02, 2015; cited 2018 20.03.2018]. Available from: https://ufm.dk/en/publications/2014/the-danish-code-of-conduct-for-research-integrity.
- [Derived] Madsen SS, Moller K, Olsen KS, Vestergaard MB, Lindberg U, Larsson HBW, Martensson J, Werner MU, Santos SAG, Asghar MS. Neuroplasticity induced by general anaesthesia: study protocol for a randomised cross-over clinical trial exploring the effects of sevoflurane and propofol on the brain - A 3-T magnetic resonance imaging study of healthy volunteers. Trials. 2020 Sep 22;21(1):805. doi: 10.1186/s13063-020-04468-y. PMID 32962743
- See also: Bigelow, Henry Jacob: Insensibility during Surgical Operations Produced by Inhalation. The Boston Medical and Surgical Journal. 1846, Volume 35, Issue 16, pp. 309-317. — http://www.nejm.org/doi/full/10.1056/NEJM184611180351601
- See also: American Society of Anesthesiologists Physical Status Classification System — https://www.asahq.org/standards-and-guidelines/asa-physical-status-classification-system
- See also: Danish Society for Anaesthesiology and Intensive Care recommendation for post-anaesthesia observation — http://www.dasaim.dk/wp-content/uploads/2019/08/Observation-efter-an%C3%A6stesi-Dec-2015.pdf
- See also: Danish Society for Anaesthesiology and Intensive Care recommendation for discharge after anaesthesia — http://www.dasaim.dk/wp-content/uploads/2019/02/udskrivningskriterier-2019.pdf
- See also: Danish Medicines Information webpage — http://pro.medicin.dk